CLINICAL TRIAL: NCT05581368
Title: Elucidating the Effects of Cannabis on Cardiovascular System
Brief Title: Studying the Effects of Cannabis on Vasculature
Acronym: SECV
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other); Canadian Cardiovascular Society (Other); Stanford University (Other); Greenstone Biosciences (Unknown)
Responsible Party: Principal Investigator, Mark Chandy, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: WCVP0001
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Inflammation; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators would like to test blood and vascular function of chronic cannabis users for signs of vascular dysfunction. The investigators e will obtain blood from a single blood draw using EDTA tubes. The investigators will separate into plasma, red blood cells, and white blood cells. The investigators will test the plasma from control and chronic cannabis users with a lipid panel, complete metabolic panel, HgbA1c, fasting glucose, and Olink inflammation panel. The investigators will retain unused plasma and peripheral blood mononuclear cells for future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Cannabis Cohort: For investigations on the effects of cannabis on the cardiovascular system, the investigators would like to recruit 50 participants with the following inclusion criteria:
  * age: 19 to 80
  * males and females
  * all ethnicities
  * cannabis use at least 3-4 times per week or more in the past 6 months (50 volunteers, experimental group)
  * no history of cardiovascular disease
  For investigations on the effects of cannabis on the cardiovascular system, the investigators will exclude cannabis users:
  * that ingest cannabis containing cannabidiol (CBD)
  * that are unable to provide a receipt for the cannabis product(s) they ingest
  * that are unwilling to stop consuming soy products and/or genistein 48 hours prior to appointments.
  Interventions: Other: Chronic Cannabis use
- Control Cohort: For investigations on the effects of cannabis on the cardiovascular system, the investigators would like to recruit 50 participants with the following inclusion criteria:
  * age: 19 to 80
  * males and females
  * all ethnicities
  * patients who do not use cannabis
  * no history of cardiovascular disease
  For investigations on the effects of cannabis on the cardiovascular system, the investigators will exclude participants:
  * that ingest cannabis
  * that are unwilling to stop consuming soy products and/or genistein 48 hours prior to appointments.

INTERVENTIONS:
Other: Chronic Cannabis use — The investigators will test levels of inflammation and vascular dysfunction in participants who chronically use cannabis.
  Groups: Chronic Cannabis Cohort

SUMMARY:
Cannabis is commonly used globally. It is associated with psychiatric problems, but the effects on the cardiovascular system are unclear. In this project, the investigators plan to study the effects of cannabis on the cardiovascular system. This will be done by using a non-invasive test to measure blood vessel function and by using blood samples to measure inflammation. As a control for this project, the investigators would like to test the blood vessel function and inflammation levels of participants who do not use cannabis. This study will provide important information on the long term cardiovascular effects of cannabis.

DETAILED DESCRIPTION:
Cannabis is the most commonly used illicit drug in the world, but the investigators do not know the long-term effects on the cardiovascular system in humans. The investigators have data from cell culture and small animal studies that cannabis is toxic to the cardiovascular system. Recently legalized in Canada, the long-term effects of cannabis use on the cardiovascular system may not be apparent for several decades. The purpose of this study is to test the effect of cannabis use on the vascular system. Using a non-invasive test of vascular function, the investigators would like to assess the effects of cannabis on chronic cannabis users. The investigators would also like to test if cannabis use by smoking and/or vaping causes adverse cardiovascular effects acutely. Lastly, the investigators would like to test blood from chronic cannabis users for inflammatory cytokines, which could further support our hypothesis that cannabis damages the cardiovascular system via inflammation.

ELIGIBILITY:
Inclusion Criteria:

* age: 19 to 80
* males and females
* all ethnicities
* cannabis use at least 3-4 times per week or more in the past 6 months (50 volunteers, experimental group)
* patients who do not use cannabis (50 volunteers, control group)
* no history of cardiovascular disease

Exclusion Criteria:

* that ingest cannabis containing cannabidiol (CBD)
* that are unable to provide a receipt for the cannabis product(s) they ingest
* that are unwilling to stop consuming soy products and/or genistein 48 hours prior to appointments.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators plan to recruit participants from the London Health Sciences Centre HIV clinic and chronic pain clinic who use cannabis for medicinal purposes.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Inflammation | Baseline measurement.
  The investigators will measure the concentration of inflammatory cytokines using an Olink for chronic cannabis users and the control group.
Endothelial function | Baseline measurement.
  The investigators will measure the reactive hyperaemia index (RHI) using an EndPAT device for both groups.

SECONDARY OUTCOMES:
Cholesterol Level | Baseline measurement.
  The investigators will measure lipid profile (total cholesterol, LDL, HDL, ratio) for both groups.
BMI | Baseline measurement.
  The investigators will measure body-mass index or both groups.
Blood pressure | Baseline measurement.
  The investigators will measure baseline blood pressure for both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- London Regional Health Science Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided